CLINICAL TRIAL: NCT06864299
Title: Study on the Safety and Efficacy of the Trans-Carotid Artery Occlusion Shunt System Combined With Introducer Sets for Cerebral Protection During Carotid Angioplasty
Brief Title: Study on the Trans-Carotid Artery Occlusion Shunt System Combined With Introducer Sets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Wecan Medical Technology Co.,Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WKP002FIM(CN)-01
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-03

CONDITIONS: Carotid Artery Stenosis; Carotid Artery Diseases
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trans-Carotid Artery Occlusion Shunt System Combined with Introducer Sets (Experimental): Device systems for the treatment of carotid artery stenosis
  Interventions: Device: Trans-Carotid Artery Occlusion Shunt System Combined with Introducer Sets

INTERVENTIONS:
Device: Trans-Carotid Artery Occlusion Shunt System Combined with Introducer Sets — To evaluate the Safety and Efficacy of the Trans-Carotid Artery Occlusion Shunt System Combined with Introducer Sets for Cerebral Protection During Carotid Angioplasty

SUMMARY:
The objective of the study is to evaluate the Safety and Efficacy of the Trans-Carotid Artery Occlusion Shunt System Combined with Introducer Sets for Cerebral Protection During Carotid Angioplasty

DETAILED DESCRIPTION:
The physician shall strictly follow the clinical study protocol and shall not deviate from or substantially change the protocol. However, in case of emergency such as immediate risk to the subjects, which needs tobe eliminated immediately, it may be reported in written form afterwards. During the course of the study,documents such as amendments to the clinical study protocol and informed consent, requests for deviation,and resumption of the suspended clinical study shall be subject to the written approval of the Ethics Committee

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with internal carotid artery stenosis, meeting at least one of the following conditions:

  * Asymptomatic carotid artery stenosis: Stenosis severity > 70%;
  * Symptomatic carotid artery stenosis: Stenosis severity > 50%, with one or more of the following symptoms occurring within 180 days prior to the procedure: transient ischemic attack (TIA), transient visual obscurations (TVO), or mild/non-disabling stroke;
* Common carotid artery diameter > 6 mm, and meets the required vascular diameter for carotid artery stenting;
* The participant or their legal guardian is able to understand the purpose of the trial, voluntarily consent to participation, sign an informed consent form, and is willing to comply with follow-up requirements as outlined in the study protocol.

Exclusion Criteria:

* Anatomical Exclusion Criteria:

  * Patients with extensive atherosclerotic plaques in the proximal common carotid artery, which hinder safe surgical manipulation;
  * Patients with lesions in the common carotid artery access area or its proximal segment;
  * Patients with the common carotid artery bifurcation located < 5 cm from the clavicular margin;
  * Patients with tandem severe stenosis or occlusion at the target lesion site;
  * Patients who have previously received stent or graft implantation in the ipsilateral carotid artery;
  * Patients with bilateral carotid artery stenosis requiring intervention on both sides;
  * Patients with acute or subacute thrombosis, arteriovenous malformations, or other abnormal vascular structures in the target lesion or adjacent regions;
  * Patients with severe calcification or tortuosity at the target lesion site, making it difficult to deliver devices to the intended location;
* Patients with concomitant severe symptomatic stenosis in other vascular territories, including intracranial or extracranial arteries;
* Patients who have experienced an ischemic stroke within the past 3 months, which may impact endpoint evaluation;
* Patients with a history of spontaneous intracranial hemorrhage within the past 12 months;
* Patients diagnosed with carotid artery dissection;
* Patients with carotid stenosis due to non-atherosclerotic causes;
* Patients with other cardiovascular conditions that may predispose to embolism, including left ventricular aneurysm, cardiomyopathy, mechanical aortic or mitral valves, infective endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma;
* Patients with central nervous system disorders, including cranial nerve impairment, which could confound endpoint evaluation (e.g., severe dementia, secondary epilepsy, etc.);
* Patients with chronic atrial fibrillation;
* Patients with paroxysmal atrial fibrillation episodes within the past 6 months or those requiring long-term anticoagulation therapy due to paroxysmal atrial fibrillation;
* Patients who have had a myocardial infarction within the last 6 months;
* Patients who have undergone or plan to undergo coronary artery bypass grafting (CABG), endovascular stenting procedures, or heart valve surgeries within 90 days prior to the procedure, which may interfere with endpoint evaluation;
* Patients with active bleeding tendencies or significant coagulation disorders;
* Patients with a history of gastrointestinal bleeding that could interfere with antiplatelet therapy;
* Patients with preoperative liver or renal dysfunction, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels exceeding 5 times the upper limit of normal, or serum creatinine (Cr) > 3.0 mg/dL (265.2 μmol/L);
* Patients with known hypersensitivity to contrast agents, anticoagulants, antiplatelet medications, or materials used in stent delivery systems (e.g., nitinol, PTFE, nylon-based polymers);
* Patients with intracranial or other malignancies;
* Patients with a life expectancy of less than 3 years;
* Women who are planning pregnancy, pregnant, or breastfeeding;
* Patients participating in another clinical trial or those who have not withdrawn or been excluded from a trial within the last 3 months of the screening period;
* Other patients who, in the investigator's opinion, are deemed unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
The composite incidence of death, stroke, and myocardial infarction within 30 days postoperatively. | Within 30 days after procedure
  Composite incidence is the rate of occurrence of a composite endpoint, which is a combination of multiple study outcomes.

SECONDARY OUTCOMES:
Immediate technical success rate | intraoperative
  Immediate technical success is defined as the complete proximal occlusion of the common carotid artery, successful establishment of an effective retrograde blood flow pathway, and the successful reconstruction of carotid blood circulation.
The incidence of stroke | pre-discharge（up to 14 days）and 30 days post-surgery
  The incidence of stroke refers to the occurrence of stroke within the follow-up time points, including hemorrhagic and ischemic strokes.
The incidence of neurological injury | Within 24 hours post-surgery and 30 days post-surgery
  The incidence of neurological injury refers to the occurrence of neurological dysfunction within the follow-up time points, including assessment of swallowing disorders, voice disorders, and facial expression muscle impairment.
The incidence of myocardial infarction | pre-discharge（up to 14 days）and 30 days post-surgery
  The incidence of myocardial infarction refers to deaths from any cause that occur within the follow-up time points.
All-cause mortality during perioperative period (from surgery to 30 days after surgery) | Intraoperatively, pre-discharge（up to 14 days）and 30 days post-surgery
  All-cause mortality Refers to deaths from any cause that occur within the follow-up time points.
Delivery system-related complications during perioperative period (from surgery to 30 days after surgery) | Intraoperatively, pre-discharge（up to 14 days）and 30 days post-surgery
  Access-related complications refer to bleeding, rebleeding, and hematoma along the delivery access route. Hematomas include surgical wound hematoma, arterial access site hematoma, and femoral venous access site hematoma.

CONTACTS AND LOCATIONS:
Overall Officials: zhong chen, Professor, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No